CLINICAL TRIAL: NCT03365947
Title: A Phase 1/2a Single Dose-Escalating Study to Evaluate the Safety, Tolerability and Pharmacokinetic Effects of ARO-HBV in Normal Adult Volunteers and Multiple Escalating Doses Evaluating Safety, Tolerability and Pharmacodynamic Effects in HBV Patients
Brief Title: Study of ARO-HBV in Normal Adult Volunteers and Patients With Hepatitis B Virus (HBV)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AROHBV1001
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Results first posted 2024-06-04 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — JNJ-56136379

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (19):
- ARO-HBV 35 mg (Experimental): Single dose of ARO-HBV 35 mg subcutaneous (sc) injection in normal healthy volunteers
  Interventions: Drug: ARO-HBV
- ARO-HBV 100 mg (Experimental): Single dose of ARO-HBV 100 mg sc injection in normal healthy volunteers
  Interventions: Drug: ARO-HBV
- ARO-HBV 200 mg (Experimental): Single dose of ARO-HBV 200 mg sc injection in normal healthy volunteers
  Interventions: Drug: ARO-HBV
- ARO-HBV 300 mg (Experimental): Single dose of ARO-HBV 300 mg sc injection in normal healthy volunteers
  Interventions: Drug: ARO-HBV
- ARO-HBV 400 mg (Experimental): Single dose of ARO-HBV 400 mg sc injection in normal healthy volunteers
  Interventions: Drug: ARO-HBV
- Placebo (Placebo Comparator): Sterile normal saline (0.9% NaCl) sc injection in normal healthy volunteers
  Interventions: Other: Sterile Normal Saline (0.9% NaCl)
- ARO-HBV 25 mg, Q28D (Experimental): ARO-HBV 25 mg sc injection every 28 days (Q28D) in participants with chronic hepatitis B
  Interventions: Drug: ARO-HBV
- ARO-HBV 50 mg Q28D (Experimental): ARO-HBV 50 mg sc injection Q28D in participants with chronic hepatitis B
  Interventions: Drug: ARO-HBV
- ARO-HBV 100 mg Q28D (Experimental): ARO-HBV 100 mg sc injection Q28D in participants with chronic hepatitis B
  Interventions: Drug: ARO-HBV
- ARO-HBV 200 mg Q28D (Experimental): ARO-HBV 200 mg sc injection Q28D in participants with chronic hepatitis B
  Interventions: Drug: ARO-HBV
- ARO-HBV 300 mg Q28D (Experimental): ARO-HBV 300 mg sc injection Q28D in participants with chronic hepatitis B
  Interventions: Drug: ARO-HBV
- ARO-HBV 400 mg Q28D (Experimental): ARO-HBV 400 mg sc injection Q28D in participants with chronic hepatitis B
  Interventions: Drug: ARO-HBV
- ARO-HBV 100 mg Q14D (Experimental): ARO-HBV 100 mg sc injection every 14 days (Q14D) in participants with chronic hepatitis B
  Interventions: Drug: ARO-HBV
- ARO-HBV 100 mg Q7D (Experimental): ARO-HBV 100 mg sc injection every 7 days (Q7D) in participants with chronic hepatitis B
  Interventions: Drug: ARO-HBV
- ARO-HBV 300 mg, Q28D, HBeAg+/ Trt Naïve (Experimental): ARO-HBV 300 mg sc injection Q28D in hepatitis B e antigen positive/treatment naïve (HBeAg+/Trt Naïve) participants with chronic hepatitis B
  Interventions: Drug: ARO-HBV
- ARO-HBV 300 mg, Q28D, HBeAg+/ NUC (Experimental): ARO-HBV 300 mg sc injection Q28D in HBeAg+/nucleotide or nucleoside analog treated (HBeAg+/NUC) participants with chronic hepatitis B
  Interventions: Drug: ARO-HBV
- ARO-HBV 200 mg, Q7D (Experimental): ARO-HBV 200 mg sc injection Q7D in participants with chronic hepatitis B
  Interventions: Drug: ARO-HBV
- ARO-HBV 300 mg, Q7D (Experimental): ARO-HBV 300 mg sc injection Q7D in participants with chronic hepatitis B
  Interventions: Drug: ARO-HBV
- ARO-HBV 200 mg Q28D + JNJ-56136379 250 mg (Experimental): ARO-HBV 200 mg sc injection Q28D plus JNJ-56136379 250 mg in participants with chronic hepatitis B
  Interventions: Drug: ARO-HBV; Drug: JNJ-56136379

INTERVENTIONS:
Drug: ARO-HBV — sc injection
  Arms: ARO-HBV 100 mg; ARO-HBV 100 mg Q14D; ARO-HBV 100 mg Q28D; ARO-HBV 100 mg Q7D; ARO-HBV 200 mg; ARO-HBV 200 mg Q28D; ARO-HBV 200 mg Q28D + JNJ-56136379 250 mg; ARO-HBV 200 mg, Q7D; ARO-HBV 25 mg, Q28D; ARO-HBV 300 mg; ARO-HBV 300 mg Q28D; ARO-HBV 300 mg, Q28D, HBeAg+/ NUC; ARO-HBV 300 mg, Q28D, HBeAg+/ Trt Naïve; ARO-HBV 300 mg, Q7D; ARO-HBV 35 mg; ARO-HBV 400 mg; ARO-HBV 400 mg Q28D; ARO-HBV 50 mg Q28D
Other: Sterile Normal Saline (0.9% NaCl) — sc injection
  Arms: Placebo
Drug: JNJ-56136379 — oral tablets
  Arms: ARO-HBV 200 mg Q28D + JNJ-56136379 250 mg

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single- and multiple-ascending doses of ARO-HBV in healthy adult volunteers and participants with hepatitis B virus (HBV).

ELIGIBILITY:
Inclusion Criteria for Parts A & B:

* Women of childbearing potential must have a negative pregnancy test, cannot be breast feeding, and must be willing to use contraception.
* Willing to provide written informed consent and comply with study requirements

Additional Inclusion Criteria for Part B:

* Diagnosis of chronic HBV infection
* Hepatitis B surface antigen (HbsAg) at screening > or = 50 IU/mL
* Liver Elastography score < or = 10.5

Exclusion Criteria:

* Clinically significant health concerns (with the exception of HBV for Patients in Part B)
* Abnormal for any clinical safety laboratory result considered clinically significant
* Regular use of alcohol within 1 month prior to screening
* Recent use of illicit drugs
* Use of an investigational agent or device within 30 days prior to dosing or current participation in an investigational study

NOTE: additional inclusion/exclusion criteria may apply, per protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (4):
  - Research Site 5, Camperdown, New South Wales
  - Research Site 4, Clayton, Victoria
  - Research Site 3, Melbourne, Victoria
  - Research Site 6, Nedlands, Western Australia
- Research Site 7, Hong Kong, Hong Kong
- New Zealand (2):
  - Research Site 1, Grafton, Auckland
  - Research Site 2, Papatoetoe, Auckland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yuen MF, Locarnini S, Lim TH, Strasser SI, Sievert W, Cheng W, Thompson AJ, Given BD, Schluep T, Hamilton J, Biermer M, Kalmeijer R, Beumont M, Lenz O, De Ridder F, Cloherty G, Ka-Ho Wong D, Schwabe C, Jackson K, Lai CL, Gish RG, Gane E. Combination treatments including the small-interfering RNA JNJ-3989 induce rapid and sometimes prolonged viral responses in patients with CHB. J Hepatol. 2022 Nov;77(5):1287-1298. doi: 10.1016/j.jhep.2022.07.010. Epub 2022 Jul 20. PMID 35870702
- [Derived] Gane E, Yuen MF, Kakuda TN, Ogawa T, Takahashi Y, Goeyvaerts N, Lonjon-Domanec I, Vaughan T, Schluep T, Hamilton J, Njumbe Ediage E, Hillewaert V, Snoeys J, Lenz O, Talloen W, Biermer M. JNJ-73763989 pharmacokinetics and safety: Liver-targeted siRNAs against hepatitis B virus, in Japanese and non-Japanese healthy adults, and combined with JNJ-56136379 and a nucleos(t)ide analogue in patients with chronic hepatitis B. Antivir Ther. 2022 Jun;27(3):13596535221093856. doi: 10.1177/13596535221093856. PMID 35695169

RESULTS

PARTICIPANT FLOW:
Groups:
- ARO-HBV 300 mg, Q28D, HBeAg+/Trt Naïve: ARO-HBV 300 mg sc injection Q28D in hepatitis B e antigen positive/treatment naïve (HBeAg+/Trt Naïve) participants with chronic hepatitis B
- ARO-HBV 300 mg, Q28D, HBeAg+/NUC: ARO-HBV 300 mg sc injection Q28D in HBeAg+/nucleotide or nucleoside analog treated (HBeAg+/NUC) participants with chronic hepatitis B
Period: Overall Study
Arm/Group | ARO-HBV 35 mg | ARO-HBV 100 mg | ARO-HBV 200 mg | ARO-HBV 300 mg | ARO-HBV 400 mg | Placebo | ARO-HBV 25 mg, Q28D | ARO-HBV 50 mg Q28D | ARO-HBV 100 mg Q28D | ARO-HBV 200 mg Q28D | ARO-HBV 300 mg Q28D | ARO-HBV 400 mg Q28D | ARO-HBV 100 mg Q14D | ARO-HBV 100 mg Q7D | ARO-HBV 300 mg, Q28D, HBeAg+/Trt Naïve | ARO-HBV 300 mg, Q28D, HBeAg+/NUC | ARO-HBV 200 mg, Q7D | ARO-HBV 300 mg, Q7D | ARO-HBV 200 mg Q28D + JNJ-56136379 250 mg
Started | 4 | 4 | 4 | 4 | 4 | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 4 | 4 | 4 | 4 | 4 | 4 | 12
Completed | 4 | 4 | 4 | 4 | 4 | 9 | 8 | 8 | 8 | 8 | 8 | 8 | 4 | 4 | 4 | 4 | 4 | 4 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ARO-HBV 25 mg Q28D: ARO-HBV 25 mg sc injection every 28 days (Q28D) in participants with chronic hepatitis B
- ARO-HBV 300 mg, Q28D, HBeAg+/Trt Naïve: ARO-HBV 300 mg sc injection Q28D in HBeAg+/Treatment Naïve (HBeAg+/Trt Naïve) participants with chronic hepatitis B
- Total: Total of all reporting groups
Arm/Group | ARO-HBV 35 mg | ARO-HBV 100 mg | ARO-HBV 200 mg | ARO-HBV 300 mg | ARO-HBV 400 mg | Placebo | ARO-HBV 25 mg Q28D | ARO-HBV 50 mg Q28D | ARO-HBV 100 mg Q28D | ARO-HBV 200 mg Q28D | ARO-HBV 300 mg Q28D | ARO-HBV 400 mg Q28D | ARO-HBV 100 mg Q14D | ARO-HBV 100 mg Q7D | ARO-HBV 300 mg, Q28D, HBeAg+/Trt Naïve | ARO-HBV 300 mg, Q28D, HBeAg+/NUC | ARO-HBV 200 mg, Q7D | ARO-HBV 300 mg, Q7D | ARO-HBV 200 mg Q28D + JNJ-56136379 250 mg | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 4 | 4 | 4 | 4 | 4 | 4 | 12 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.0 (3.01) | 23.5 (0.67) | 24.8 (4.23) | 28.1 (8.15) | 23.6 (3.73) | 27.2 (9.08) | 42.8 (7.17) | 47.8 (6.97) | 50.8 (12.48) | 47.5 (6.75) | 52.1 (7.42) | 41.0 (9.91) | 48.9 (7.71) | 40.7 (6.59) | 31.8 (7.90) | 36.0 (4.93) | 53.2 (6.67) | 50.7 (12.39) | 44.9 (9.19) | 40.3 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 3 | 2 | 6 | 3 | 2 | 2 | 3 | 0 | 2 | 1 | 1 | 2 | 2 | 3 | 1 | 4 | 42
  Male | 2 | 2 | 3 | 1 | 2 | 4 | 5 | 6 | 6 | 5 | 8 | 6 | 3 | 3 | 2 | 2 | 1 | 3 | 8 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 1 | 0 | 0 | 1 | 6 | 6 | 8 | 8 | 5 | 6 | 3 | 1 | 3 | 4 | 4 | 3 | 12 | 74
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 13
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
  White | 3 | 0 | 3 | 3 | 3 | 8 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Possibly or Probably Related to Treatment
Description: An adverse event (AE) is any untoward medical occurrence which does not necessarily have to have a causal relationship with this treatment. TEAEs were defined as AEs with onset after administration of the study drug, or when a preexisting medical condition increases in severity or frequency after study drug administration. Assessment of causality utilized 3 possible categories: not related, possibly related and probably related.
Time Frame: NHV participants: up to Day 29 (± 2 days); CHB participants: Day 113 (± 2 days)
Population: Safety Population: all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- ARO-HBV 35 mg: Single dose of ARO-HBV 35 mg sc injection in normal healthy volunteers
- ARO-HBV 25 mg Q28D: ARO-HBV 25 mg sc injection every 28 days (Q28D) in participants with chronic hepatitis B (CHB)
Arm/Group | ARO-HBV 35 mg | ARO-HBV 100 mg | ARO-HBV 200 mg | ARO-HBV 300 mg | ARO-HBV 400 mg | Placebo | ARO-HBV 25 mg Q28D | ARO-HBV 50 mg Q28D | ARO-HBV 100 mg Q28D | ARO-HBV 200 mg Q28D | ARO-HBV 300 mg Q28D | ARO-HBV 400 mg Q28D | ARO-HBV 100 mg Q14D | ARO-HBV 100 mg Q7D | ARO-HBV 300 mg, Q28D, HBeAg+/Trt Naïve | ARO-HBV 300 mg, Q28D, HBeAg+/NUC | ARO-HBV 200 mg, Q7D | ARO-HBV 300 mg, Q7D | ARO-HBV 200 mg Q28D + JNJ-56136379 250 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 4 | 4 | 4 | 4 | 4 | 4 | 12
Participants
  Possibly Related TEAE | 1 | 1 | 1 | 1 | 1 | 5 | 2 | 2 | 1 | 1 | 5 | 3 | 0 | 2 | 2 | 0 | 0 | 0 | 0
  Probably Related TEAE | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 2 | 1 | 0 | 2 | 0

2. Secondary Outcome: Part A, Pharmacokinetics (PK) of ARO-HBV Analytes: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Day 1: 0 (pre-dose), 15 minutes, 0.5, 1, 2, 3, 6, 24 & 48 hours post-dose
Population: PK Population: All NHV participants receiving ARO-HBV (participants receiving placebo were excluded from the analysis per statistical analysis plan [SAP]). Participants with a valid assessment.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ARO-HBV 35 mg | ARO-HBV 100 mg | ARO-HBV 200 mg | ARO-HBV 300 mg | ARO-HBV 400 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 4
ng/mL
  Analyte: JNJ-73763976 | 160 (106) | 536 (390) | 1320 (331) | 2920 (1670) | 4280 (1340)
  Analyte: JNJ-73763924 | 43.0 (25.8) | 117 (45.2) | 363 (89.5) | 827 (447) | 1010 (398)

3. Secondary Outcome: Part A, PK of ARO-HBV Analytes : Time to Maximum Plasma Concentration (Tmax)
Time Frame: Day 1: 0 (pre-dose), 15 minutes, 0.5, 1, 2, 3, 6, 24 & 48 hours post-dose
Population: PK Population: All NHV participants receiving ARO-HBV (participants receiving placebo were excluded from the analysis per SAP). Participants with a valid assessment.
Measure: Median (Full Range); unit: hours
Arm/Group | ARO-HBV 35 mg | ARO-HBV 100 mg | ARO-HBV 200 mg | ARO-HBV 300 mg | ARO-HBV 400 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 4
hours
  Analyte: JNJ-73763976 | 6.00 [6.00 to 6.03] | 6.00 [3.00 to 6.00] | 6.00 [2.00 to 6.00] | 6.03 [2.00 to 6.05] | 6.00 [6.00 to 6.00]
  Analyte: JNJ-73763924 | 6.00 [2.00 to 6.00] | 6.00 [2.00 to 6.00] | 1.50 [0.500 to 6.00] | 2.02 [1.00 to 3.00] | 6.00 [6.00 to 6.00]

4. Secondary Outcome: Part A, PK of ARO-HBV Analytes: Area Under the Plasma Concentration Versus Time Curve From Zero to 24 Hours (AUC0-24)
Time Frame: Day 1: 0 (pre-dose), 15 minutes, 0.5, 1, 2, 3, 6, 24 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | ARO-HBV 35 mg | ARO-HBV 100 mg | ARO-HBV 200 mg | ARO-HBV 300 mg | ARO-HBV 400 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 4
h*ng/mL
  Analyte: JNJ-76763976 | 1830 (1190) | 5480 (2540) | 17800 (4180) | 35500 (17200) | 44600 (15100)
  Analyte: JNJ-76763924: number analyzed (Participants) | 1 | 4 | 4 | 4 | 4
  Analyte: JNJ-76763924 | 327 (NA) — 1 participant analyzed | 1250 (330) | 4320 (965) | 8140 (3160) | 9720 (3680)

5. Secondary Outcome: Part A, PK of ARO-HBV Analytes: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUCinf)
Time Frame: Day 1: 0 (pre-dose), 15 minutes, 0.5, 1, 2, 3, 6, 24 & 48 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | ARO-HBV 35 mg | ARO-HBV 100 mg | ARO-HBV 200 mg | ARO-HBV 300 mg | ARO-HBV 400 mg
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 0
h*ng/mL
  Analyte: JNJ-6763976: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Analyte: JNJ-6763976 |  | 5820 (NA) — 1 participant analyzed | 12600 (NA) — 1 participant analyzed | 14800 (NA) — 1 participant analyzed |
  Analyte: JNJ-76763924 | 365 (NA) — 1 participant analyzed | 1530 (NA) — 1 participant analyzed | 4610 (1190) | 8170 (3420) |

6. Secondary Outcome: Part A, PK of ARO-HBV Analytes: Area Under the Plasma Concentration Versus Time Curve From Zero to the Time of the Last Quantifiable Concentration (AUC0-t)
Time Frame: Day 1: 0 (pre-dose), 15 minutes, 0.5, 1, 2, 3, 6, 24 & 48 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | ARO-HBV 35 mg | ARO-HBV 100 mg | ARO-HBV 200 mg | ARO-HBV 300 mg | ARO-HBV 400 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 4
h*ng/mL
  Analyte: JNJ-76763976 | 1830 (1190) | 5740 (2480) | 20100 (5250) | 37900 (16900) | 46900 (17400)
  Analyte: JNJ-76763924 | 254 (127) | 1250 (330) | 4600 (1130) | 8330 (2820) | 9940 (3990)

7. Secondary Outcome: Part A, PK of ARO-HBV Analytes: Terminal Elimination Half-Life (t½)
Time Frame: Day 1: 0 (pre-dose), 15 minutes, 0.5, 1, 2, 3, 6, 24 & 48 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ARO-HBV 35 mg | ARO-HBV 100 mg | ARO-HBV 200 mg | ARO-HBV 300 mg | ARO-HBV 400 mg
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 0
hours
  Analyte: JNJ-6763976: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Analyte: JNJ-6763976 |  | 6.45 (NA) — 1 participant analyzed | 5.83 (NA) — 1 participant analyzed | 9.16 (NA) — 1 participant analyzed |
  Analyte: JNJ-76763924 | 7.52 (NA) — 1 participant analyzed | 5.97 (NA) — 1 participant analyzed | 6.48 (1.23) | 6.02 (2.34) |

8. Secondary Outcome: Part A, PK of ARO-HBV Analytes: Dose-Normalized AUC0-24
Time Frame: Day 1: 0 (pre-dose), 15 minutes, 0.5, 1, 2, 3, 6, 24 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*ng/mL/mg
Arm/Group | ARO-HBV 35 mg | ARO-HBV 100 mg | ARO-HBV 200 mg | ARO-HBV 300 mg | ARO-HBV 400 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 4
h*ng/mL/mg
  Analyte: NJ-76763976 | 52.1 (34.1) | 54.8 (25.4) | 88.9 (20.9) | 118 (57.3) | 111 (37.7)
  Analyte: JNJ-6763924: number analyzed (Participants) | 1 | 4 | 4 | 4 | 4
  Analyte: JNJ-6763924 | 9.34 (NA) — 1 participant analyzed | 12.5 (3.30) | 21.6 (4.83) | 27.1 (10.5) | 24.3 (9.20)

9. Secondary Outcome: Part A, PK of ARO-HBV Analytes: Dose-Normalized AUC0-t
Time Frame: Day 1: 0 (pre-dose), 15 minutes, 0.5, 1, 2, 3, 6, 24 & 48 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*ng/mL/mg
Arm/Group | ARO-HBV 35 mg | ARO-HBV 100 mg | ARO-HBV 200 mg | ARO-HBV 300 mg | ARO-HBV 400 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 4
h*ng/mL/mg
  Analyte: JNJ-6763976 | 52.1 (34.1) | 57.4 (24.8) | 101 (26.3) | 126 (56.5) | 117 (43.5)
  Analyte:JNJ-76763924 | 7.25 (3.63) | 12.5 (3.30) | 23.0 (5.65) | 27.8 (9.39) | 24.8 (9.98)

10. Secondary Outcome: Part A, PK of ARO-HBV Analytes: Dose-Normalized Cmax
Time Frame: Day 1: 0 (pre-dose), 15 minutes, 0.5, 1, 2, 3, 6, 24 & 48 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | ARO-HBV 35 mg | ARO-HBV 100 mg | ARO-HBV 200 mg | ARO-HBV 300 mg | ARO-HBV 400 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 4
ng/mL/mg
  Analyte: JNJ-76763976 | 4.56 (3.03) | 5.36 (3.90) | 6.58 (1.65) | 9.72 (5.58) | 10.7 (3.34)
  Analyte: JNJ-76763924 | 1.23 (0.737) | 1.17 (0.452) | 1.81 (0.448) | 2.76 (1.49) | 2.53 (0.994)

11. Secondary Outcome: Change From Baseline in HBV Surface Antigen (HBsAg) From Day 1 Pre-Dose Baseline to Post-Dose Nadir in Participants Chronically Infected With HBV
Time Frame: Part B (multiple-ascending dose [MAD] phase) only: up to 113 days
Population: Pharmacodynamic (PD) Population: participants who received at least one dose of study treatment and had PD assessment from baseline and assessment from post-baseline.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | ARO-HBV 25 mg Q28D | ARO-HBV 50 mg Q28D | ARO-HBV 100 mg Q28D | ARO-HBV 200 mg Q28D | ARO-HBV 300 mg Q28D | ARO-HBV 400 mg Q28D | ARO-HBV 100 mg Q14D | ARO-HBV 100 mg Q7D | ARO-HBV 300 mg, Q28D, HBeAg+/Trt Naïve | ARO-HBV 300 mg, Q28D, HBeAg+/NUC | ARO-HBV 200 mg, Q7D | ARO-HBV 300 mg, Q7D | ARO-HBV 200 mg Q28D + JNJ-56136379 250 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 4 | 4 | 4 | 4 | 4 | 4 | 12
IU/mL | -1.083 (0.5320) | -1.199 (0.2525) | -1.695 (0.4921) | -1.769 (0.4018) | -1.534 (0.3080) | -1.889 (0.6948) | -1.549 (0.2956) | -1.412 (0.4153) | -2.252 (1.0177) | -2.492 (0.6493) | -2.316 (0.6979) | -1.879 (0.2676) | -1.687 (0.3887)

ADVERSE EVENTS:
Time Frame: From the screening period (Day -60) and up to the end of the follow-up of the study (Day 398)
Arm/Group | ARO-HBV 35 mg | ARO-HBV 100 mg | ARO-HBV 200 mg | ARO-HBV 300 mg | ARO-HBV 400 mg | Placebo | ARO-HBV 25 mg Q28D | ARO-HBV 50 mg Q28D | ARO-HBV 100 mg Q28D | ARO-HBV 200 mg Q28D | ARO-HBV 300 mg Q28D | ARO-HBV 400 mg Q28D | ARO-HBV 100 mg Q14D | ARO-HBV 100 mg Q7D | ARO-HBV 300 mg, Q28D, HBeAg+/Trt Naïve | ARO-HBV 300 mg, Q28D, HBeAg+/NUC | ARO-HBV 200 mg, Q7D | ARO-HBV 300 mg, Q7D | ARO-HBV 200 mg Q28D + JNJ-56136379 250 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/10 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/10 | 0/8 | 0/8 | 1/8 | 0/8 | 0/8 | 1/8 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 1/4 | 1/12
Other Adverse Events (participants affected / at risk) | 1/4 | 4/4 | 3/4 | 3/4 | 3/4 | 8/10 | 6/8 | 6/8 | 5/8 | 4/8 | 6/8 | 7/8 | 3/4 | 4/4 | 3/4 | 2/4 | 4/4 | 3/4 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARO-HBV 35 mg (N=4) | ARO-HBV 100 mg (N=4) | ARO-HBV 200 mg (N=4) | ARO-HBV 300 mg (N=4) | ARO-HBV 400 mg (N=4) | Placebo (N=10) | ARO-HBV 25 mg Q28D (N=8) | ARO-HBV 50 mg Q28D (N=8) | ARO-HBV 100 mg Q28D (N=8) | ARO-HBV 200 mg Q28D (N=8) | ARO-HBV 300 mg Q28D (N=8) | ARO-HBV 400 mg Q28D (N=8) | ARO-HBV 100 mg Q14D (N=4) | ARO-HBV 100 mg Q7D (N=4) | ARO-HBV 300 mg, Q28D, HBeAg+/Trt Naïve (N=4) | ARO-HBV 300 mg, Q28D, HBeAg+/NUC (N=4) | ARO-HBV 200 mg, Q7D (N=4) | ARO-HBV 300 mg, Q7D (N=4) | ARO-HBV 200 mg Q28D + JNJ-56136379 250 mg (N=12)
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retroperitoneal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARO-HBV 35 mg (N=4) | ARO-HBV 100 mg (N=4) | ARO-HBV 200 mg (N=4) | ARO-HBV 300 mg (N=4) | ARO-HBV 400 mg (N=4) | Placebo (N=10) | ARO-HBV 25 mg Q28D (N=8) | ARO-HBV 50 mg Q28D (N=8) | ARO-HBV 100 mg Q28D (N=8) | ARO-HBV 200 mg Q28D (N=8) | ARO-HBV 300 mg Q28D (N=8) | ARO-HBV 400 mg Q28D (N=8) | ARO-HBV 100 mg Q14D (N=4) | ARO-HBV 100 mg Q7D (N=4) | ARO-HBV 300 mg, Q28D, HBeAg+/Trt Naïve (N=4) | ARO-HBV 300 mg, Q28D, HBeAg+/NUC (N=4) | ARO-HBV 200 mg, Q7D (N=4) | ARO-HBV 300 mg, Q7D (N=4) | ARO-HBV 200 mg Q28D + JNJ-56136379 250 mg (N=12)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ill-defined disorder (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 3 | 0 | 3 | 2 | 4 | 1 | 1 | 1 | 1 | 3 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular access site bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular access site inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular access site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site bruise (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 1 | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral hyperaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site discolouration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Posterior capsule opacification (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Crystal urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis C antibody positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Ear swelling (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperparathyroidism primary (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retroperitoneal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor retains first right to publish results for this multi-center study, and thereafter can review results communications prior to release and can embargo communications regarding trial results for a period that is 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication of results but can require removal of its confidential information (excluding results).

DOCUMENTS (2):
  • Study Protocol (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT03365947/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-03): https://cdn.clinicaltrials.gov/large-docs/47/NCT03365947/SAP_002.pdf